CLINICAL TRIAL: NCT05018793
Title: Safety of Cultured Autologous Adult Adipose Derived Mesenchymal Stem Cell Versus Cultured Allogeneic Adult Umbilical-cord Derived Mesenchymal Stem Cell Intrathecal Injection for the Treatment of Spinal Cord Injury
Brief Title: Safety of Cultured Autologous Adult Adipose Derived Mesenchymal Stem Cell Versus Cultured Allogeneic Adult Umbilical-cord Derived Mesenchymal Stem Cell Intrathecal Injection for SCI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SC-8-GR-10-02
Record Dates: First submitted 2021-08-19; First posted 2021-08-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; SCI; stem cell treatment
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Single intrathecal injection of 100 million cells
  Interventions: Biological: autologous adipose derived mesenchymal stem cells; Biological: AlloRx

INTERVENTIONS:
Biological: autologous adipose derived mesenchymal stem cells — cultured autologous adult adipose derived mesenchymal stem cells
Biological: AlloRx — Cultured Allogeneic Adult Umbilical-cord Derived Mesenchymal Stem Cell Intrathecal injection for

SUMMARY:
This trial will study the safety and efficacy of intrathecal injection of cultured autologous adult adipose derived mesenchymal stem cells versus cultured allogeneic adult umbilical-cord derived mesenchymal stem cells for the treatment of spinal cord injury

DETAILED DESCRIPTION:
Studies have shown that stem cell treatment is safe and efficacious for the treatment of spinal cord injury (SCI). This patient funded trial aims to study the safety and efficacy of intrathecal injection of cultured autologous adult adipose derived mesenchymal stem cells (AD-MSCs) versus cultured allogeneic adult umbilical-cord derived mesenchymal stem cell for the treatment of SCI. Patients with SCI will receive a single intrathecal injection of AD-MSCs. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Spinal Cord Injury
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Anticoagulation medicine use
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Previous organ transplant
* Hypersensitivity to sulfur
* Continued drug abuse
* Pre-menopausal women not using contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

SECONDARY OUTCOMES:
Efficacy: American Spinal Injury Association Impairment Scale (ASIA) | Four year follow-up
  It will be completed for each follow up point

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Athens Beverly Hills Medical Group, Glyfada, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bydon M, Dietz AB, Goncalves S, Moinuddin FM, Alvi MA, Goyal A, Yolcu Y, Hunt CL, Garlanger KL, Del Fabro AS, Reeves RK, Terzic A, Windebank AJ, Qu W. CELLTOP Clinical Trial: First Report From a Phase 1 Trial of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells in the Treatment of Paralysis Due to Traumatic Spinal Cord Injury. Mayo Clin Proc. 2020 Feb;95(2):406-414. doi: 10.1016/j.mayocp.2019.10.008. Epub 2019 Nov 27. PMID 31785831
- [Background] Hur JW, Cho TH, Park DH, Lee JB, Park JY, Chung YG. Intrathecal transplantation of autologous adipose-derived mesenchymal stem cells for treating spinal cord injury: A human trial. J Spinal Cord Med. 2016 Nov;39(6):655-664. doi: 10.1179/2045772315Y.0000000048. Epub 2015 Jul 24. PMID 26208177
- [Background] Roberts TT, Leonard GR, Cepela DJ. Classifications In Brief: American Spinal Injury Association (ASIA) Impairment Scale. Clin Orthop Relat Res. 2017 May;475(5):1499-1504. doi: 10.1007/s11999-016-5133-4. Epub 2016 Nov 4. No abstract available. PMID 27815685